CLINICAL TRIAL: NCT00770081
Title: A 28-week Extension to a 24-week Multicenter, Randomized, Double-blind, Active-controlled Clinical Trial to Evaluate the Safety and Tolerability of Vildagliptin (50 mg qd) Versus Sitagliptin (25 mg qd) in Patients With Type 2 Diabetes and Severe Renal Insufficiency
Brief Title: Safety and Tolerability of Vildagliptin Versus Sitagliptin in Patients With Type 2 Diabetes and Severe Renal Insufficiency (28-week Extension Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237A23138E1
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2; Renal Insufficiency
Keywords: Type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — Vildagliptin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 50mg qd vildagliptin
  Interventions: Drug: vildagliptin
- 2 (Active Comparator): sitagliptin (25mg qd)
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: vildagliptin — 50mg qd
  Arms: 1
Drug: sitagliptin — 25mg qd
  Arms: 2

SUMMARY:
This clinical trial is designed to provide additional information on the safety and tolerability of vildagliptin (50 mg once daily (qd)) and sitagliptin (25 mg qd) when used in patients with type 2 diabetes mellitus(T2DM) and severe renal insufficiency (Glomerular filtration rate (GFR) < 30 mL/min) for a period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Complete the core study and consent for extension

Exclusion Criteria:

* Patient unable to comply with core study requirements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Assessment of treatment emergent adverse events (including hypoglycemia events and other events of special interest) | 52 weeks

SECONDARY OUTCOMES:
To assess hemoglobin A1c (HbA1c) and fasting plasma glucose (FPG) reduction from baseline after 52 weeks of treatment | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (86):
- United States (86):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Anasazi Internal Medicine, Phoenix, Arizona
  - Sonoran Health Specialists, Scottsdale, Arizona
  - Mary K. Richards, MD. PA, Little Rock, Arkansas
  - University of Arkanasas for Medical Sciences, Little Rock, Arkansas
  - Burlingame, California
  - John Muir Clinical Research, Concord, California
  - Academic Medical Research Institute, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Northern California Institute for Bone Health, Oakland, California
  - Dr. Wei Feng, Pasadena, California
  - Sierra Clinical Research - Orangevale, Roseville, California
  - California Institute of Renal Research, San Diego, California
  - Denver Nephrology PC, Denver, Colorado
  - Western Nephrology & Metabolic Bone Disease PC, Lakewood, Colorado
  - Western Nephrology & Metabolic Bone Disease PC, Westminster, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Nephrology Associates of South Miami, Aventura, Florida
  - University of Florida Shands Hospital, Gainesville, Florida
  - Center for Diabetes & Endocrine Care, Hollywood, Florida
  - Larry Levinson, D.O., PA, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Osler Medical Clinical Research, Melbourne, Florida
  - Tampa Bay Nephrology Associates, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Boise Kidney & Hypertension Institiute, Meridian, Idaho
  - Iowa Diabetes & Endocrinology Research Center PLC, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa
  - Cray Diabetes Education Center, Kansas City, Kansas
  - Cotton-O'Neil Diabetes & Endocrinology Center, Topeka, Kansas
  - Metabolic Center of Louisiana, Baton Rouge, Louisiana
  - Dolby Research, LLC, Baton Rouge, Louisiana
  - Bruce Samuels LLC, Covington, Louisiana
  - Egan Healthcare, Metairie, Louisiana
  - Crescent City Clinical Research Center, Metairie, Louisiana
  - Arthritis and Diabetes Clinic, Monroe, Louisiana
  - Northwest Louisiana Nephrology Research, Shreveport, Louisiana
  - Joslin Diabetes Center at North Arundel Hospital, Glen Burnie, Maryland
  - Biolab Research, LLC, Rockville, Maryland
  - Harvard University (Joslin Diabetes Center), Boston, Massachusetts
  - Genesys Integrated Group Practice, PC, Flint, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Phillips Medical Services, PLLC, Jackson, Mississippi
  - Mississippi Medical Research, LLC, Picayune, Mississippi
  - Diabetes and Endocrinology Specialist, Inc, Chesterfield, Missouri
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Arms, Dodge, Robinson, Wilber & Crouch, Inc., Kansas City, Missouri
  - Washington U School of Medicine, St Louis, Missouri
  - Platte Valley Medical Group, Kearney, Nebraska
  - Creighton Diabetes Center, Omaha, Nebraska
  - Creighton Nephrology, Omaha, Nebraska
  - UMDNJ-Robert Wood Johnson, New Brunswick, New Jersey
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - Downstate University of Brooklyn, Brooklyn, New York
  - HRRG, Orchard Park, New York
  - SUNY - Upstate Medical University, Syracuse, New York
  - Meritcare Medical Group, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Hightop Medical Research Center, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Portland Hypertension and Nephrology, Oregon City, Oregon
  - Lehigh Valley Hospital-Dept. of Medicine Research, Allentown, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Renal Endocrine Associates, P. C., Pittsburgh, Pennsylvania
  - Aiken Center for Clinical Research, Aiken, South Carolina
  - Medical U of South Carolina, Charleston, South Carolina
  - SC Nephrology and Hyptertension Center, Inc., Orangeburg, South Carolina
  - Sumter Medical Specialists, Sumter, South Carolina
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - Medical Nephrology Associates, Dyersburg, Tennessee
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Baylor Clinic (BCM 621), Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Renal Associates, P.A., San Antonio, Texas
  - Allied Institute of Medicine, San Antonio, Texas
  - Central Utah Clinic, American Fork, Utah
  - Clinical Research and Consulting Center, LLC, Fairfax, Virginia
  - Nephrology Associates of Northern Virginia, Fairfax, Virginia
  - Medical College of Virginia, Richmond, Virginia
  - Washington State University at Spokane, Spokane, Washington
  - UW Health - West Clinic, Madison, Wisconsin

REFERENCES:
- See also: Results for CLAF237A23138E1 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5923